CLINICAL TRIAL: NCT01481766
Title: Optimizing Early Child Development in the Primary Care Practice Setting: Pragmatic Randomized Trial of Iron Treatment for Young Children With Non-anemic Iron Deficiency (OptEC)
Brief Title: Iron Treatment for Young Children With Non-anemic Iron Deficiency
Acronym: OptEC
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: The Hospital for Sick Children (Other)
Collaborators: Canadian Institutes of Health Research (CIHR) (Other Government); Mead Johnson Nutrition (Industry); Mount Sinai Hospital, Canada (Other); Unity Health Toronto (Other)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Quadruple | Purpose: Treatment
Other Study IDs: 1000027782
Record Dates: First submitted 2011-11-22; First posted 2011-11-30 (Estimated); Results first posted 2025-10-30 (Actual); Last update posted 2025-10-30 (Actual); Status verified 2025-10

CONDITIONS: Non-anemic Iron Deficiency
Keywords: child development; screening; Non-anemic iron deficiency; primary care pediatrics; prevention and health promotion
MeSH Terms: conditions — Iron Deficiencies | interventions — ferrous sulfate; Nutrition Assessment

STUDY DESIGN:
Who Masked: Participant, Care Provider, Investigator, Outcomes Assessor
Masking Description: The research pharmacy prepared ferrous sulfate and placebo in bottles of similar appearance and weight. The placebo was developed by the research pharmacy, was similar in color and consistency to the active agent, and had a distinctive taste.
  Individuals masked to group allocation throughout the study included parents, attending physicians, research assistants, study personnel conducting outcome assessments, data analysts, and investigators. The biostatistician was unmasked after completion of data collection and locking of the database. The principal investigator was unmasked after the analysis.
Oversight: Data Monitoring Committee: No

ARMS (4):
- Iron plus dietary counseling (Non-anemic iron deficiency) (Experimental)
  Interventions: Dietary Supplement: Ferrous Sulfate; Behavioral: Dietary counseling
- Placebo plus dietary counseling (Non-anemic iron deficiency) (Placebo Comparator)
  Interventions: Dietary Supplement: Placebo; Behavioral: Dietary counseling
- Iron sufficient (No Intervention): From the screening cohort of it is anticipated that 25 children will have iron deficiency anemia and an equal number of randomly selected children with iron sufficiency (n=25) will be sampled. These children will be compared to the children with non-anemic iron deficiency.
- Iron deficiency anemia (Active Comparator): From the screening cohort of it is anticipated that 25 children will have iron deficiency anemia and an equal number of randomly selected children with iron sufficiency (n=25) will be sampled. These children will be compared to the children with non-anemic iron deficiency.
  Interventions: Dietary Supplement: Ferrous Sulfate; Behavioral: Dietary counseling

INTERVENTIONS:
Dietary Supplement: Ferrous Sulfate — 6 mg elemental iron/kg/day (0.4 ml/kg/day) in 2 or 3 divided doses (at the discretion of prescribing study doctor) for four months plus dietary counseling
  Other Names: Brand name: Fer-In-Sol by Mead Johnson Nutrition; NPN #: 00762954
  Arms: Iron deficiency anemia; Iron plus dietary counseling (Non-anemic iron deficiency)
Dietary Supplement: Placebo — 0.4 ml/kg/day in 2 or 3 divided doses (at the discretion of prescribing study doctor) for four months plus dietary counseling
  Arms: Placebo plus dietary counseling (Non-anemic iron deficiency)
Behavioral: Dietary counseling — Dietary counseling will include written recommendations regarding maximum daily cow's milk intake, varied solid food intake including high iron containing foods, and avoidance of foods which reduce iron absorption.
  Arms: Iron deficiency anemia; Iron plus dietary counseling (Non-anemic iron deficiency); Placebo plus dietary counseling (Non-anemic iron deficiency)

SUMMARY:
The pre-school years are critical years for children to acquire early learning skills such as language, fine motor and social skills; this is termed early child development. Primary care doctors (family doctors and pediatricians) are in a unique position to identify children with health or developmental problems. Screening is the process of testing healthy people for the earliest signs of health problems, followed by treatment, with the expectation that screening will improve the health of those screened. The focus of this research is screening young children for the earliest signs of iron deficiency (low blood iron levels) followed by treatment with oral iron.

Previous research has shown that children with later stages of iron deficiency have serious delays in their development. Some research has shown that these delays may persist into young adulthood often with a significant reduction in intelligence. Early stages of iron deficiency may be difficult for parents or doctors to detect, and a blood test is usually needed. However, Canadian guidelines do not recommend screening all children for iron deficiency, because there is not enough good quality research to prove that screening is effective.

In this study, the investigators will ask parents to allow their child between the ages of 1 to 3 years to have a blood test for iron levels. If the blood level is low, the child will be randomly assigned to receive either oral iron liquid for 4 months plus diet counseling, or a placebo liquid plus diet counseling. A psychologist will measure each child's early learning ability before and after the treatment. If this approach to screening children's blood iron levels followed by treatment improves children's development, parents and doctors may consider that routine blood screening tests are justified. Overall, this research is an important step to improving the ways in which primary care doctors can ensure that children have the best start to life-long health and achievement.

ELIGIBILITY:
Inclusion Criteria:

* Age between 12 and 40 months attending any well child visit
* Informed parental consent

Exclusion Criteria:

* developmental disorder
* genetic, chromosomal or syndromic condition
* chronic medical condition (with the exception of asthma and allergies)
* chronic anemia, iron deficiency, or recent oral iron supplementation or treatment
* prematurity, with a gestational age of less than 35 weeks
* low birth weight less than 2,500 g;
* attending the office for an acute illness, such as a viral illness, or other health concern other than for a well-child assessment
* any contraindications to receiving elemental iron
* the use of any natural health product containing the same medicinal ingredient(s) as the investigational product
* English is not spoken to the child in the home or in a child care setting
* CRP level ≥10 mg/L

Ages: 12 Months to 40 Months | Sex: All | Healthy Volunteers: Yes
Age Groups: Child
Enrollment: 127 (Actual)
Dates: Start 2012-06 (Actual); Primary Completion 2018-10 (Actual); Study Completion 2018-12 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Parkin C Parkin, MD, Principal Investigator — The Hospital for Sick Children
Locations (2):
- Canada (2):
  - St. Michael's Hospital, Toronto, Ontario
  - The Hospital for Sick Children, Toronto, Ontario

REFERENCES:
- [Result] Parkin PC, Borkhoff CM, Macarthur C, Abdullah K, Birken CS, Fehlings D, Koroshegyi C, Maguire JL, Mamak E, Mamdani M, Thorpe KE, Zlotkin SH, Zuo F; TARGet Kids! Collaboration. Randomized Trial of Oral Iron and Diet Advice versus Diet Advice Alone in Young Children with Nonanemic Iron Deficiency. J Pediatr. 2021 Jun;233:233-240.e1. doi: 10.1016/j.jpeds.2021.01.073. Epub 2021 Feb 4. PMID 33548262
- [Result] Gingoyon A, Borkhoff CM, Koroshegyi C, Mamak E, Birken CS, Maguire JL, Fehlings D, Macarthur C, Parkin PC. Chronic Iron Deficiency and Cognitive Function in Early Childhood. Pediatrics. 2022 Dec 1;150(6):e2021055926. doi: 10.1542/peds.2021-055926. PMID 36412051
- [Derived] Parkin PC, Koroshegyi C, Mamak E, Borkhoff CM, Birken CS, Maguire JL, Thorpe KE; TARGet Kids! Collaboration. Association between Serum Ferritin and Cognitive Function in Early Childhood. J Pediatr. 2020 Feb;217:189-191.e2. doi: 10.1016/j.jpeds.2019.09.051. Epub 2019 Nov 2. PMID 31685227
- [Derived] Abdullah K, Thorpe KE, Mamak E, Maguire JL, Birken CS, Fehlings D, Hanley AJ, Macarthur C, Zlotkin SH, Parkin PC. An internal pilot study for a randomized trial aimed at evaluating the effectiveness of iron interventions in children with non-anemic iron deficiency: the OptEC trial. Trials. 2015 Jul 14;16:303. doi: 10.1186/s13063-015-0829-4. PMID 26170014
- [Derived] Abdullah K, Thorpe KE, Mamak E, Maguire JL, Birken CS, Fehlings D, Hanley AJ, Macarthur C, Zlotkin SH, Parkin PC. Optimizing early child development for young children with non-anemic iron deficiency in the primary care practice setting (OptEC): study protocol for a randomized controlled trial. Trials. 2015 Apr 2;16:132. doi: 10.1186/s13063-015-0635-z. PMID 25873050

RESULTS

PARTICIPANT FLOW:
Recruitment Details: Healthy children were enrolled while attending a scheduled health supervision visit at 1 of 8 primary care practices participating in a primary care research network called TARGet Kids! in Toronto, Canada. Enrollment began on June 15, 2012, and data collection was completed on November 9, 2018.
Pre-assignment Details: 220 children were assessed for eligibility. Based on each child's baseline blood tests (hemoglobin and ferritin), children with nonanemic iron deficiency (NAID) were eligible for the randomized trial; and children with iron deficiency anemia (IDA) and iron sufficiency (IS) were eligible for the open label study (not randomized). Therefore, 60 children were eligible for the randomized arms; 67 children were eligible for the open label study (not randomized). The total enrolled was 127 children.
Groups:
- Non-anemic iron deficiency - randomized to ferrous sulfate plus diet advice: liquid ferrous sulfate (6 mg elemental iron/kg/d, Fer-In-Sol, supplied by Mead Johnson Nutrition) in 2 divided doses daily by mouth for 4 months plus diet advice (parents received a written guide, developed by the investigators, for improving iron status including recommendations on iron-containing foods, foods that increase and inhibit iron absorption, and feeding practices that may prevent iron deficiency)
- Non-anemic iron deficiency randomized to placebo plus diet advice: liquid placebo in 2 divided doses daily by mouth for 4 months plus diet advice (parents received a written guide, developed by the investigators, for improving iron status including recommendations on iron-containing foods, foods that increase and inhibit iron absorption, and feeding practices that may prevent iron deficiency)
- Iron sufficient - not randomized: Normal hemoglobin and normal ferritin. No treatment.
- Iron deficiency anemia - not randomized: Low hemoglobin and low ferritin. Received oral iron and diet advice for 4 months
Period: 4 months
Arm/Group | Non-anemic iron deficiency - randomized to ferrous sulfate plus diet advice | Non-anemic iron deficiency randomized to placebo plus diet advice | Iron sufficient - not randomized | Iron deficiency anemia - not randomized
Started | 31 | 29 | 30 | 37
Completed | 28 | 27 | 29 | 32
Not Completed | 3 | 2 | 1 | 5
Not completed — Lost to Follow-up | 3 | 2 | 1 | 5
Period: 12 months
Arm/Group | Non-anemic iron deficiency - randomized to ferrous sulfate plus diet advice | Non-anemic iron deficiency randomized to placebo plus diet advice | Iron sufficient - not randomized | Iron deficiency anemia - not randomized
Started | 28 | 27 | 29 | 32
Completed | 21 | 19 | 24 | 29
Not Completed | 7 | 8 | 5 | 3
Not completed — Lost to Follow-up | 7 | 8 | 5 | 3

BASELINE CHARACTERISTICS:
Groups:
- NAID - Iron Plus Diet Advice: From the screening cohort, children with NAID (nonanemic iron deficiency) were invited to participate in an RCT. This group was randomized to receive Ferrous Sulfate 6 mg elemental iron/kg/day in 2 divided doses for four months plus diet advice
- NAID - Placebo Plus Diet Advice: From the screening cohort, children with NAID (nonanemic iron deficiency) were invited to participate in an RCT. This group was randomized to receive Placebo in 2 divided doses for four months plus diet advice
- IS - Iron Sufficient: From the screening cohort, a random sample of children with Iron Sufficiency were invited to participate in a prospective observational arm. They received diet advice only.
- IDA - Iron Deficiency Anemia: From the screening cohort, children with Iron Deficiency Anemia (IDA) were invited to participate in a prospective observational arm. They received usual care, including Ferrous Sulfate 6 mg elemental iron/kg/day in 2 divided doses for four months plus diet advice.
- Total: Total of all reporting groups
Arm/Group | NAID - Iron Plus Diet Advice | NAID - Placebo Plus Diet Advice | IS - Iron Sufficient | IDA - Iron Deficiency Anemia | Total
Number analyzed (Participants) | 31 | 29 | 30 | 37 | 127
Age, Categorical [Count of Participants; unit: Participants]
  <=18 years | 31 | 29 | 30 | 37 | 127
  Between 18 and 65 years | 0 | 0 | 0 | 0 | 0
  >=65 years | 0 | 0 | 0 | 0 | 0
Age, Continuous [Mean (Standard Deviation); unit: months] | 24.0 (8.1) | 24.5 (6.6) | 27.97 (8.70) | 20.32 (6.13) | 23.97 (7.32)
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 13 | 17 | 15 | 19 | 64
  Male | 18 | 12 | 15 | 18 | 63
Race/Ethnicity, Customized [Count of Participants; unit: Participants]
  Maternal Ethnicity: other European | 14 | 21 | 20 | 19 | 74
  Maternal Ethnicity: Other | 17 | 8 | 10 | 18 | 53
Region of Enrollment [Number; unit: participants]
  Canada | 31 | 29 | 30 | 37 | 127
Early Learning Composite (ELC) [Mean (Standard Deviation); unit: points] — ELC is a measure of infant cognition (similar to IQ). In populations, infants have a mean score of 100 points and standard deviation of 15 points. A higher score indicates higher cognitive ability. Four cognitive skills are summarized into an Early Learning Composite score - Fine Motor, Visual Reception, Receptive Language, and Expressive Language.
  points | 108.7 (15.2) | 109.2 (14.9) | 106.33 (10.55) | 103.73 (12.82) | 106.81 (13.26)
Serum Ferritin [Mean (Standard Deviation); unit: ug/L] | 9.7 (2.3) | 10.1 (2.5) | 26.63 (10.84) | 7.14 (3.22) | 13.04 (4.63)

OUTCOME MEASURES:

1. Primary Outcome: Early Learning Composite (ELC) From the Mullen Scales of Early Learning
Description: ELC is a measure of infant cognition (similar to IQ). In populations, infants have a mean score of 100 points and standard deviation of 15 points. A higher score indicates higher cognitive ability. Four cognitive skills are summarized into an Early Learning Composite score - Fine Motor, Visual Reception, Receptive Language, and Expressive Language.
Time Frame: Baseline and 4 months after enrollment
Population: ELC 4 months after enrollment
Measure: Mean (Standard Deviation); unit: units on a scale
Groups:
- NAID - ferrous sulfate plus diet advice; Iron deficiency anemia: Ferrous sulfate plus diet advice
- NAID - placebo plus diet advice: Placebo plus diet advice
- Iron sufficient: Diet advice only
Arm/Group | NAID - ferrous sulfate plus diet advice | NAID - placebo plus diet advice | Iron sufficient | Iron deficiency anemia
Number analyzed (Participants) | 28 | 27 | 29 | 32
units on a scale | 113.0 (19.3) | 113.5 (12.6) | 110.48 (10.16) | 107.94 (13.69)

2. Secondary Outcome: Serum Ferritin
Description: Blood samples analyzed for serum ferritin
Time Frame: 4 months after enrollment
Measure: Mean (Standard Deviation); unit: ug/L
Arm/Group | NAID - ferrous sulfate plus diet advice | NAID - placebo plus diet advice | Iron sufficient | Iron deficiency anemia
Number analyzed (Participants) | 28 | 27 | 30 | 33
ug/L | 37.8 (30.8) | 20.4 (11.2) | 27.13 (9.06) | 57.55 (40.44)

ADVERSE EVENTS:
Time Frame: 4 months
Arm/Group | NAID - Iron plus diet advice | NAID - Placebo plus diet advice | IS - Iron sufficient | IDA - Iron deficiency anemia
All-Cause Mortality (participants affected / at risk) | 0/28 | 0/27 | 0/29 | 0/32
Serious Adverse Events (participants affected / at risk) | 0/28 | 0/27 | 0/29 | 0/32
Other Adverse Events (participants affected / at risk) | 16/28 | 7/27 | 0/29 | 16/32
OTHER ADVERSE EVENTS; cells are participants affected of the arm's N at risk (number of events):
Term (organ system) | NAID - Iron plus diet advice (N=28) | NAID - Placebo plus diet advice (N=27) | IS - Iron sufficient (N=29) | IDA - Iron deficiency anemia (N=32)
Change in stool (Gastrointestinal disorders) | 16 (16) | 7 (7) | 0 (0) | 16 (16) — Constipation, Black stool, loose stool

LIMITATIONS AND CAVEATS:
For children with NAID enrolled in the RCT, limitations include: our study population with high maternal education; our end points may not have been long enough; we were not able to measure chronicity of iron deficiency; the effect estimate for our primary outcome was based on findings from previous iron studies, but there is uncertainty regarding what is considered a meaningful treatment effect

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: Yes

DOCUMENTS (1):
  • Study Protocol and Statistical Analysis Plan (2012-02-11): https://cdn.clinicaltrials.gov/large-docs/66/NCT01481766/Prot_SAP_000.pdf